CLINICAL TRIAL: NCT03354312
Title: Multicenter, Randomized, Split-mouth Study to Evaluate the Acceptance and Preference of Lidocaine Gel Compared to Injection Anesthesia After Non Surgical Periodontal Treatment
Brief Title: Acceptance and Preference of Lidocaine Gel Compared to Injection Anesthesia After Non Surgical Periodontal Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chemische Fabrik Kreussler & CO GmbH (Industry)
Collaborators: Anfomed GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: DyMZIS-01
Record Dates: First submitted 2017-11-14; First posted 2017-11-27 (Actual); Last update posted 2018-12-20 (Actual); Status verified 2018-12

CONDITIONS: Periodontitis
Keywords: scaling and root planing; topical anesthesia
MeSH Terms: conditions — Periodontitis | interventions — Lidocaine; Gels; Carticaine; Epinephrine

STUDY DESIGN:
Intervention Model Description: The randomization determines if a subject will be assigned to receive either lidocaine gel or articaine injection anesthesia as the first anesthesia during SRP Treatment of the right upper and lower jaw. The second anesthesia during SRP at visit 2 will be carried out with the remaining anesthetic on the left side of the upper and lower jaw.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lidocaine/Articaine (Experimental): Lidocaine Hydrochloride 1% Gel anesthesia / Articaine hydrochloride/epinephrine (adrenaline) hydrochloride anesthesia
  Interventions: Drug: Lidocaine Hydrochloride 1% Gel; Drug: Articaine hydrochloride/epinephrine (adrenaline) hydrochloride
- Articaine/Lidocaine (Experimental): Articaine hydrochloride/epinephrine (adrenaline) hydrochloride anesthesia / Lidocaine Hydrochloride 1% Gel anesthesia
  Interventions: Drug: Lidocaine Hydrochloride 1% Gel; Drug: Articaine hydrochloride/epinephrine (adrenaline) hydrochloride

INTERVENTIONS:
Drug: Lidocaine Hydrochloride 1% Gel — Cylinder vials with 1.7 g gel containing 34 mg lidocaine (1 g gel contains 20 mg lidocaine) will be used. Application of the gel into the periodontal pockets or the sulcus according to summary of product characteristics (SmPC). A total dose of 40 mg lidocaine should not be exceeded.
  Other Names: Dynexan Mundgel®
Drug: Articaine hydrochloride/epinephrine (adrenaline) hydrochloride — Cylinder vials with 1.7 ml solution for injection containing 68 mg articaine and 0.0102 mg epinephrine (1 ml contains 40 mg articaine and 0.006 mg epinephrine) will be used. Infiltration anesthesia for the upper jaw and infiltration or nerve block anesthesia for the lower jaw with articaine solution for injection according to SmPC. Adults can be treated with up to 7 mg articaine per kg of body weight per treatment session.
  Other Names: Ultracain® D-S 1:200,000

SUMMARY:
This project is a national, open label, multicenter, randomized split-mouth study in patients from 18 to 70 years of age to compare the efficacy and acceptability of lidocaine gel compared to injection anesthesia with articaine (infiltration anesthesia for the upper jaw and infiltration or nerve block anesthesia for the lower jaw). It is planned that about 90 patients with a proven moderate periodontitis will be enrolled in 5 German study centers.

Dynexan Mundgel® (lidocaine hydrochloride) is a topical anesthetic gel containing lidocaine that is commercially available as an anesthetic for temporary, symptomatic treatment of pain at the oral mucosa, gingiva and lips. The gold standard for scaling and root planing (SRP) is still the use of injection anesthesia. This raises the question what kind of anesthesia patients would prefer if they had a free choice.

For this study Ultracaine® D-S 1:200,000 (articaine hydrochloride/epinephrine hydrochloride) was selected as the injectable comparator drug because it is the most frequently used anesthetic drug for infiltration and nerve-block anesthesia in Germany at present.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent must be available
* Willingness and ability to comply with scheduled visits, treatment plan, and other study procedures
* Patient systemically healthy except for controlled diabetes and hypertension
* Patients with comparable periodontal status of the right and left jaw, with ≥ 3 teeth with pockets ≥ 4 mm and ≤ 7 mm per quadrant
* Female patients of childbearing potential must practice highly effective contraception methods

Exclusion Criteria:

* Generalized severe periodontitis with pockets > 8 mm
* More than 2 pockets > 7 mm and ≤ 8 mm per quadrant
* Contraindicated for treatment with the investigational product, the comparator drug, or meet warnings and precautions for use specifications in accordance with the approved SmPCs as follows:

  * Hypersensitivity to the investigational product, the comparator drug or to any of their respective excipients
  * Hypersensitivity to other local anesthetics of the amide type
  * Severe uncontrolled and untreated excitation and conduction disorder of the heart
  * Acute decompensated heart failure
  * Severe renal or hepatic disease/dysfunction
  * Untreated or uncontrolled diabetes type 2
  * Severe hypertension and severe hypotension
  * Narrow-angle glaucoma
  * Hyperthyroidism
  * Paroxysmal tachycardia or high-frequency absolute arrhythmia
  * Myocardial infarction within the last 6 months
  * Coronary artery bypass within the last 3 months
  * Concurrent use of non-cardio selective beta blockers (e.g. propranolol)
  * Pheochromocytoma
  * Concurrent treatment with tri-cyclic antidepressants or monoamine oxidase (MAO) inhibitors
* Use of painkillers or anti-inflammatory drugs 24 hours before the first treatment
* Antibiotic prophylaxis or treatment with antibiotics
* Use of any anxiolytic medication
* Periodontal treatment within the last 3 months
* Continuing orthodontic treatment
* Concurrent use of another investigational medication
* Participation in another clinical trial within the last 3 months
* Women who are pregnant or breastfeeding, or planning pregnancy while enrolled in the study
* Persons who are in a dependency or working relationship with the sponsor or investigator
* A subject who, in the opinion of the investigator will be uncooperative or unable to comply with study procedures

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2017-12-05 (Actual); Primary Completion 2018-11-02 (Actual); Study Completion 2018-11-02 (Actual)

PRIMARY OUTCOMES:
Acceptance and preference of topical lidocaine mouth gel anesthesia | 1 hour post-dose of second treatment
  To compare acceptance and preference of topical lidocaine mouth gel anesthesia vs. injection anesthesia with articaine in patients undergoing subgingival debridement by comparing the proportion of patients after the second periodontal treatment who prefer topical anesthesia with lidocaine gel against the injection anesthesia with articaine to a proportion of 0.5; the patient rates the preferred anesthesia method on a questionnaire by stating if the patient's preference is treatment with anesthetic gel, treatment with anesthetic injection, or no preference

SECONDARY OUTCOMES:
Assessment of pain | 1 hour post-dose
  Comparative assessment of pain the patients experienced during treatment; a visual analogue scale (100mm, 0 = no pain, 100 = maximum pain) will be used for maximum pain and average pain Rating after each treatment visit
Side Effects | 1, 5, 25 hours post-dose
  Evaluate type and number of side effects (incl. after-effects due to study Treatment up to 24h after each treatment visit by use of a patient diary)
Handling/Application | 1 hour post-dose
  Compare the handling/application of both methods; the treating physician rates the handling/application on a questionnaire by using German school grades (1 = very good, 2 = good, 3 = satisfactory, 4 = adequate, 5 = inadequate, 6 = insufficient) after each treatment visit.
Onset of anesthetic effect | 1 hour post-dose
  Compare the onset of anesthetic effect in both treatment groups; the treating physician rates the onset of the anesthetic effect on a questionnaire by using German school grades (1 = very good, 2 = good, 3 = satisfactory, 4 = adequate, 5 = inadequate, 6 = insufficient) after each treatment visit.
Duration of anesthetic effect | 1 hour post-dose
  Compare the duration of anesthetic effect in both treatment groups; the treating physician rates the duration of the anesthetic effect on a questionnaire by using German school grades (1 = very good, 2 = good, 3 = satisfactory, 4 = adequate, 5 = inadequate, 6 = insufficient) after each treatment visit.
Patient compliance | 1 hour post-dose
  Compare the patient compliance in both treatment groups; the treating physician rates the patient compliance on a questionnaire by using German school grades (1 = very good, 2 = good, 3 = satisfactory, 4 = adequate, 5 = inadequate, 6 = insufficient) after each treatment visit.
Treating physicians preference | 1 hour post-dose of second treatment
  Evaluation which of the anesthetic methods the treating physician prefers. The treating physician rates the preferred anesthesia method on a questionnaire by stating if the treating physician's preference is treatment with anesthetic gel, treatment with anesthetic injection, or no preference
Anesthesia re-application/rescue anesthesia | 1 hour post-dose
  Assess the number of re-application of the anesthetic gel or the rescue anesthesia injections that are required in every treatment group
Overall patient satisfaction with anesthesia | 1 hour post-dose
  Evaluation of the overall patient satisfaction with anesthesia. The patient rates the overall satisfaction on a questionnaire by using German school grades (1 = very good, 2 = good, 3 = satisfactory, 4 = adequate, 5 = inadequate, 6 = insufficient) after each treatment visit.
Willingness to pay | 1 hour post-dose of second treatment
  Evaluation of the willingness to pay for lidocaine gel by using a questionnaire (willingness to pay 0, 1-5, 5-10, 10-15, 15-20 or >20 €)
Re-Evaluation of patients preference | 25 hours post-dose of second treatment
  Re-evaluation of preference of topical lidocaine mouth gel anesthesia vs. injection anesthesia with articaine 24 h after end of last treatment. The patient again rates the preferred anesthesia method by stating if his/her preference is treatment with anesthetic gel, treatment with anesthetic injection, or no preference. The preference 24 h after end of last treatment is collected by using the patient diary.

CONTACTS AND LOCATIONS:
Locations (5):
- Germany (5):
  - Praxis Dr. Heckel, Röttenbach, Bavaria
  - Praxis Dr. Petersilka, Würzburg, Bavaria
  - Universitätsklinikum Giessen und Marburg GmbH, Standort Marburg, Marburg, Hesse
  - Universitätsklinikum Schleswig-Holstein, Klinik für Zahnerhaltungskunde und Parodontologie, Kiel, Schleswig-Holstein
  - Charité - Universitätsmedizin Berlin Charité Centrum Zahn-, Mund- und Kieferheilkunde CC 3, Berlin